CLINICAL TRIAL: NCT00000863
Title: A Phase II Study of WR 6026 for Pneumocystis Carinii Pneumonia in People With HIV Infection
Brief Title: A Study of WR 6026 in the Treatment of Pneumocystis Carinii Pneumonia (PCP) in HIV-Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 314; 11289 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Administration, Oral; WR 6026
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; AIDS-Related Opportunistic Infections | interventions — 8-aminoquinoline

INTERVENTIONS:
Drug: Sitamaquine

SUMMARY:
To evaluate the efficacy of WR 6026 once daily in the treatment of mild PCP. To evaluate the safety and tolerance of WR 6026. To assess the correlation between plasma WR 6026 concentrations and outcome/toxicity.

DETAILED DESCRIPTION:
All patients will receive an initial loading dose of WR 6026, followed the next morning and each morning thereafter by 1 of 2 lower doses of WR 6026 taken in a fasting state for 3 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Any medications not listed as excluded will be permitted on study.

[ AS PER AMENDMENT 4/11/97:PCP prophylaxis is permitted if initiated after the Day 21 evaluation has been completed.]

Patients must have:

* Documented HIV infection.
* Documented PCP.
* On a room air ABG, the PO2 value greater than or equal to 70 mm Hg and the (A-a) DO2 less than 35 mm Hg.
* Signed informed consent from parent or legal guardian for those patients less than 18 years of age.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Known hypersensitivity to quinolines.
* If patient is unwilling or unable to discontinue other medications with anti-PCP activity during the treatment period of this study.

Concurrent Medication:

Excluded:

* Any patient unwilling or unable to discontinue other medications with anti-PCP activity during the treatment period of this study (e.g., TMP/SMX, sulfonamides, dapsone, pentamidine, trimetrexate, atovaquone, clindamycin, azithromycin, pyrimethamine, primaquine).
* Methemoglobinemia-producing agents (dapsone, primaquine, sulfonamides, chloroquine, nitrofurantoin, nitrates and nitrites).

Patients with the following prior conditions or symptoms are excluded:

* History of G6PD deficiency, hemoglobin M abnormality, or NAD methemoglobin reductase deficiency.

Prior Medication:

Excluded:

* More than 24 hours receipt of anti-PCP treatment for the current episode of PCP. Receipt of prior PCP prophylaxis is permitted, as long as it is discontinued at study entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45
Dates: Study Completion 1998-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dohn M, Study Chair; Petty B, Study Chair; Black J, Study Chair; Frame P, Study Chair
Locations (12):
- United States (12):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - Queens Med. Ctr., Honolulu, Hawaii
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Weiss Memorial Hosp., Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Indiana Univ. School of Medicine, Wishard Memorial, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio

REFERENCES:
- [Background] Petty BG, Black JR, Hendrix CW, Lewis LD, Basiakos Y, Feinberg J, Pattison DG, Hafner R. Escalating multiple-dose safety and tolerance study of oral WR 6026 in HIV-infected subjects: AIDS clinical trials group 173. J Acquir Immune Defic Syndr. 1999 May 1;21(1):26-32. doi: 10.1097/00126334-199905010-00004. PMID 10235511